CLINICAL TRIAL: NCT01307241
Title: Evaluation of RFC Transporter & MTHFR SNP's, as Well as hEN1 and DCK Expression as Prognostic Factors in Patients With Acute Lymphoblastic Leukemia.
Brief Title: RFC and MTHFR SNPs & hENT1- dCK Expression as Prognostic Factors in ALL & hENT1- dCK Expression as Prognostic Factors in AML
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute of Cancerología (Other Government)
Responsible Party: Principal Investigator, DR. MYRNA CANDELARIA, Clinical researcher., National Institute of Cancerología
Other Study IDs: 010/020/ICI
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Acute Lymphoblastic Leukemia.; Acute Myeloblastic Leukemia
Keywords: Acute lymphoblastic leukemia; prognostic factor; pharmacogenetics.
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- one cohort: Adult patients with ALL attending at the Instituto Nacional de Cancerologia Mexico.

SUMMARY:
Results of actual treatment in ALL are not optimal. New prognostic factors, which may determine clinical & molecular response are required. Hyper-CVAD is an internationally accepted schema for such patients. The objective of this pilot study is to evaluate polymorphisms regarding RFC (reduced folate carrier) and MTHFR enzyme, which may affect the function of these proteins, and therefore the intracellular bioavailability of methotrexate. Also, the expression levels of hENT1 and dCK will be evaluated, since such genes codify for citarabine intracellular transport and activation, respectively. Clinical characteristics will be tabulated and analyzed for responders & non-responders patients. Uni- & multivariate analysis will be done to evaluate factors influencing on response and survival.

ELIGIBILITY:
Inclusion Criteria:

* Age: older than 15 years.
* Male, female.
* Normal renal & liver functions.
* Without previous treatment.
* Candidate to be treated with hyperCVAD Schema (ALL patients).
* Candidate to receive induction remission with cytarabine (AML patients)

Exclusion Criteria:

* Patients not candidate to receive methotrexate or cytarabine.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate clinical response | December 2012
  To evaluate clinical response after ending Hyper-CVAD schema for ALL patients. To evaluate clinical response & DFS in relation with hENT1 & dCK expression levels in AML patients.
Clinical responses in relation with SNP's or gene expression | clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: myrna candelaria, md, Principal Investigator — Instituto Nacional de Cancerología Mexico
Locations (1):
- Instituto Nacional de Cancerologia, Mexico City, Mexico City, Mexico